CLINICAL TRIAL: NCT07248644
Title: Immunosuppressant Discontinuation in Elderly Patients With Ulcerative Colitis And Long-term Remission
Brief Title: Discontinuation of Thiopurine Therapy in Elderly Patients With Ulcerative Colitis
Acronym: IDEA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEA
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: thiopurines; 5-ASA; mesalazine
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Discontinuation Arm (Experimental): Immediate cessation of thiopurine therapy while continuing standard mesalamine
  Interventions: Drug: Discontinuation of thiopurines.
- Continuation Arm (No Intervention): Maintenance of current thiopurine dose together with mesalamine.

INTERVENTIONS:
Drug: Discontinuation of thiopurines. — Because thiopurine-related toxicity rises with age while late-onset UC tends to be less aggressive, replacing thiopurines with high-dose oral mesalazine (≥ 3 g/day) may preserve remission and simultaneously reduce long-term oncological and infectious risks.
  Arms: Discontinuation Arm

SUMMARY:
IDEA is a Phase IV, prospective, randomised, open-label, multicentre clinical trial designed to evaluate the safety and efficacy of withdrawing thiopurines in elderly (≥60 years) patients with ulcerative colitis (UC) who are in sustained clinical and biological remission. The study compares discontinuation of thiopurines versus continuation while maintaining background mesalamine therapy over 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥60 years at screening.
2. Established diagnosis of ulcerative colitis according to ECCO criteria.
3. Clinical and endoscopic remission ≥12 months (Mayo score ≤2, subscore ≤1) according to clinical practice.
4. Treatment with a thiopurine (azathioprine 1-2.5 mg/kg/day or mercaptopurine 0.75-1.5 mg/kg/day) for ≥60 months. Treatment at stable doses (minimum effective dose without adverse events in the last 12 months.
5. In case of concomitant treatment with oral mesalazine, the dose must´ve been stable for ≥12 months.
6. Clinical remission (at the discretion of the investigator) for at least 3 years, without the need for treatment with oral or intravenous steroids or biological agents (topical rectal treatments are permitted as well as oral mesalazine if the dose has remained stable over the past 12 months).
7. Colonoscopy performed within 6 months prior to the start of the study in endoscopic remission (Mayo endoscopic index 0) according to clinical practice.
8. Two consecutive (centralised determinations in the period of one month) basal faecal calprotectin values <150 mg/kg during screening.
9. Written informed consent.

Exclusion Criteria:

1. Ulcerative proctitis (maximum observed extension <25 cm throughout the course of the disease)
2. History of colectomy or imminent need for surgery.
3. Presence of ileoanal reservoir
4. History of complex perianal disease
5. Intolerance to oral 5-ASA treatment
6. Previous or concomitant biologic anti-TNF (vedolizumab, Ustekinumab) or JAK-inhibitor therapy for any condition.
7. Severe chronic renal insufficiency, defined as serum creatinine ≥ 2 mg/dL (estimated glomerular filtration rate ≤ 30 mL/min/1.73 m²).
8. Abnormal hepatic laboratory parameters, defined as AST, ALT, alkaline phosphatase, or GGT > 2X the upper limit of normal (ULN) at screening.
9. Hematologic abnormalities at screening, defined as any of the following: absolute neutrophil count < 1,500 cells/mm³, lymphocytes < 500 cells/mm³, platelets < 120,000 cells/mm³, or haemoglobin < 12 g/dL (females) / < 13 g/dL (males).
10. Any condition that in the investigator's opinion may compromise study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Biologic Relapse at 24 Months in Elderly UC Patients After Thiopurine Discontinuation | From enrollment to the end of treatment suspension at 24 months.
  To compare the biological-relapse rate at 24 months in elderly patients with quiescent ulcerative colitis (UC) in long-term remission who discontinue thiopurines versus those who continue thiopurine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Margalida Calafat, MD, PhD, Principal Investigator — Spanish Working Group on Crohn's disease and ulcerative colitis (GETECCU)